CLINICAL TRIAL: NCT05044078
Title: Effects of Autogenic and Reciprocal Inhibition Techniques With Conventional Therapy in Mechanical Neck Pain- A Randomized Control Trial
Brief Title: Effects of Autogenic and Reciprocal Inhibition Techniques With Conventional Therapy in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Mahrukh Siddiqi, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSiddiqi
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Mechanical Neck Pain
Keywords: Neck Pain; Manual Therapies; Therapy-Soft Tissue; Muscle Stretching exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: It is a randomized control trial. Total 80 patients will be recruited, 40 in each group that includes 10 patients as a dropout in both groups. There will be one interventional group and one active comparator group. Treatment will be allocated using a random number sheet generated by statistician. Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor involved in the clinical trial will be prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Autogenic Inhibition) (Experimental): Autogenic Inhibition (5 reps, 10-sec hold, 5-sec rest in between each rep, 1 set, in all sessions) will be provided with the Conventional therapy including neck Isometric strengthening exercise (Neck Flexion, Extension, Both sides Rotation, and Neck Bending with each 5 rep, 10-sec hold, 1 set, in all sessions), Maitland Central posterio-anterior glide (Grade 1 and 2, 30 rep, 3 sets, in all sessions) and hot pack (10 minutes in all sessions on the back of the neck)
  Interventions: Other: Autogenic Inhibition MET
- Group 2 (Reciprocal Inhibition) (Active Comparator): Reciprocal Inhibition (5 reps, 10-sec hold, 5-sec rest in between each rep, 1 set, in all sessions) will be provided with the with same Conventional therapy as in group 1 .
  Interventions: Other: Reciprocal Inhibition MET

INTERVENTIONS:
Other: Autogenic Inhibition MET — If a sub-maximal contraction of the muscle is followed by stretching of the same muscle it is known as Autogenic Inhibition MET.
  Arms: Group 1 (Autogenic Inhibition)
Other: Reciprocal Inhibition MET — If a submaximal contraction of a muscle is followed by stretching of the opposite muscle then this is known as Reciprocal Inhibition MET.
  Arms: Group 2 (Reciprocal Inhibition)

SUMMARY:
The objective of this randomized control trial is to determine the effectiveness of Autogenic and Reciprocal Inhibition techniques with conventional therapy in mechanical neck pain to improve Pain, Range of Motion, and Functional Disability in long term. This study is being conducted at the Physiotherapy department of Sindh Institute of Physical Medicine and Rehabilitation, Karachi (former institute of Dow University of Health Sciences) among 80 patients with mechanical neck pain on the basis of non-probability purposive sample technique with screening for study criteria through a consultant physician (blinded) . After taking informed consent all participants will be randomly allocated in two groups through second researcher who is not involved in screening, baseline assessment and providing intervention. Group 1 will receive Autogenic Inhibition muscle energy technique (MET) with conventional therapy and Group 2 will receive Reciprocal inhibition MET with conventional therapy. A total of 12 sessions will be provided. Outcomes will be assessed at baseline, after 1st session, and at last session.

ELIGIBILITY:
Inclusion Criteria:

* Moderate intensity (3.5-7.4cm) Pain on VAS
* Limited or Painful Cervical ROM
* Pain more than 4 weeks (sub-acute and chronic)
* 20-50 years Age

Exclusion Criteria:

* Any Symptom and sign of Radiculopathy and Myelopathy
* Any neurological disease like Multiple Sclerosis, Parkinson or Stroke
* Taking any Pain medication
* Trigger Point of Upper Trapezius
* Any fracture, surgical procedure, or trauma of the cervical spine
* Any red flag or signs of serious pathology like rheumatic or inflammatory diseases, malignancy, infection, or vascular disease such as Vertebro-Basilar Insufficiency.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the 10 centimetre Visual analogue scale (VAS-10cm) at first day. | Baseline and 1 day
  The patient will asked to mark the pain Intensity on the line of 0-10cm that measures the level of pain. The 0 refers no pain and 10-cm refers excruciating pain as perceived as maximum.
Change from baseline in pain on the 10 centimetre Visual analogue scale (VAS-10cm) at 12 session. | Baseline and 3 weeks
  The patient will asked to mark the pain Intensity on the line of 0-10cm that measures the level of pain. The 0 refers no pain and 10-cm refers excruciating pain as perceived as maximum
Change from baseline in disability on the Neck Disability Index (NDI) at first session. | Baseline and 1 day
  This questionnaire has been designed to give information as to neck pain of patient has affected the ability to manage in everyday life. Patient will be asked to answer every section and mark in each section only the one box that most closely describes his or her problem. The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score.The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. The 0 points or 0% means : no activity limitations, 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability. It is available in both English and Urdu. Minimum Detectable Change (90% confidence): 5 points or 10% points.
Change from baseline in disability on the Neck Disability Index (NDI) at 12 sessions. | Baseline and 3 weeks
  This questionnaire has been designed to give information as to neck pain of patient has affected the ability to manage in everyday life. Patient will be asked to answer every section and mark in each section only the one box that most closely describes his or her problem. The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score.The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. The 0 points or 0% means : no activity limitations, 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability. It is available in both English and Urdu. Minimum Detectable Change (90% confidence): 5 points or 10% points.
Change from baseline in Neck range of motion measured through Goniometer at first session. | Baseline and 1 day
  It is an instrument that is used to measures the available Range of Motion around a joint in degrees. The investigator will appropriately place goniometer to measure the range of motions of neck (Flexion, extension, right and left lateral flexion and rotation). Lower the reading of goniometer suggests decreased in range of motion and vice versa.
Change from baseline in Neck range of motion measured through Goniometer at 12 session. | Baseline and 3 weeks
  It is an instrument that is used to measures the available Range of Motion around a joint in degrees. The investigator will appropriately place goniometer to measure the range of motions of neck (Flexion, extension, right and left lateral flexion and rotation). Lower the reading of goniometer suggests decreased in range of motion and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Mahrukh Siddiqi, MSAPT, Principal Investigator — Dow University of Health Sciences; Saeed Akhter, MSPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Pakistan; Aftab Ahmed Mirza Baig, MSAPT, Principal Investigator — Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Pakistan.
Locations (1):
- Sindh Institue of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Safiri S, Kolahi AA, Hoy D, Buchbinder R, Mansournia MA, Bettampadi D, Ashrafi-Asgarabad A, Almasi-Hashiani A, Smith E, Sepidarkish M, Cross M, Qorbani M, Moradi-Lakeh M, Woolf AD, March L, Collins G, Ferreira ML. Global, regional, and national burden of neck pain in the general population, 1990-2017: systematic analysis of the Global Burden of Disease Study 2017. BMJ. 2020 Mar 26;368:m791. doi: 10.1136/bmj.m791. PMID 32217608
- [Background] Binder AI. Neck pain. BMJ Clin Evid. 2008 Aug 4;2008:1103. PMID 19445809
- [Background] Evans G. Identifying and treating the causes of neck pain. Med Clin North Am. 2014 May;98(3):645-61. doi: 10.1016/j.mcna.2014.01.015. Epub 2014 Mar 22. PMID 24758966
- [Background] Heintz MM, Hegedus EJ. Multimodal management of mechanical neck pain using a treatment based classification system. J Man Manip Ther. 2008;16(4):217-24. doi: 10.1179/106698108790818260. PMID 19771194
- [Background] Karnath BM. Identifying the musculoskeletal causes of neck pain [Internet]. Rheumatologynethreefiverk.com. [cited 2021 Apr 2]. Available from: https://www.rheumatologynetwork.com/view/identifying-musculoskeletal-causes-neck-pain
- [Background] Binder AI. Cervical spondylosis and neck pain. BMJ. 2007 Mar 10;334(7592):527-31. doi: 10.1136/bmj.39127.608299.80. No abstract available. PMID 17347239
- [Background] Miller J, Gross A, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL. Manual therapy and exercise for neck pain: a systematic review. Man Ther. 2010 Aug;15(4):334-54. PMID 20593537
- [Background] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Background] What can you do about non-specific neck pain? Institute for Quality and Efficiency in Health Care (IQWiG); 2019.
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- [Background] Waxenbaum JA, Woo MJ, Lu M. Physiology, Muscle Energy. 2024 Jan 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559029/ PMID 32644455
- [Background] Elsevier. Muscle Energy Techniques E-Book [Internet]. Elsevier.com. [cited 2021 Apr 2]. Available from: https://www.elsevier.com/books/muscle-energy-techniques-with-dvdrom/chaitow/978-0-7020-3243-1.
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Osama M, Shakil Ur Rehman S. Effects of static stretching as compared to autogenic inhibition and reciprocal inhibition muscle energy techniques in the management of mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 May;70(5):786-790. doi: 10.5455/JPMA.9596. PMID 32400728
- [Background] Howell ER. The association between neck pain, the Neck Disability Index and cervical ranges of motion: a narrative review. J Can Chiropr Assoc. 2011 Sep;55(3):211-21. PMID 21886283
- [Background] Gandbhir VN, Cunha B. Goniometer. 2020 Jun 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558985/ PMID 32644411
- [Background] Kahl C, Cleland JA. Visual analogue scale, numeric pain rating scale and the McGill pain Questionnaire: an overview of psychometric properties. Phys Ther Rev. 2005;10(2):123-8
- [Background] Thomas E, Cavallaro AR, Mani D, Bianco A, Palma A. The efficacy of muscle energy techniques in symptomatic and asymptomatic subjects: a systematic review. Chiropr Man Therap. 2019 Aug 27;27:35. doi: 10.1186/s12998-019-0258-7. eCollection 2019. PMID 31462989
- [Background] Gross AR, Kay T, Hondras M, Goldsmith C, Haines T, Peloso P, Kennedy C, Hoving J. Manual therapy for mechanical neck disorders: a systematic review. Man Ther. 2002 Aug;7(3):131-49. doi: 10.1054/math.2002.0465. PMID 12372310
- [Background] Satria Nugraha MH, Antari NKAJ, Saraswati NLPGK. The efficacy of muscle energy technique in individuals with mechanical neck pain: A systematic review. Sport Fit J. 2020;8(2):91.
- [Background] Yadav H. Efficacy of Muscle Energy Technique and Deep Neck Flexors Training in Mechanical Neck Pain: A Randomized Clinical trial. Int J Ther Rehabil. 2014;4(1).
- [Background] Jalal Y, Ahmad A, Rahman AU; Irfanullah; Daud M; Aneela. Effectiveness of muscle energy technique on cervical range of motion and pain. J Pak Med Assoc. 2018 May;68(5):811-813. PMID 29885191
- [Background] Osama M, Tassadaq N, Malik RJ. Effect of muscle energy techniques and facet joint mobilization on spinal curvature in patients with mechanical neck pain: A pilot study. J Pak Med Assoc. 2020 Feb;70(2):344-347. doi: 10.5455/JPMA.14189. PMID 32063632
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Background] Branco. Cervical Range of Motion and Isometrics [Internet]. Prpaspinesurgery.com. [cited 2021 Apr 4]. Available from: https://www.prpaspinesurgery.com/wpcontent/uploads/Isometrics-cervical.pdf.
- [Background] Cervical Spine Goniometry [Internet]. Uwa.edu. [cited 2021 Apr 2]. Available from: http://at.uwa.edu/gon/cspine.htm
- [Background] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Background] Ackelman BH, Lindgren U. Validity and reliability of a modified version of the neck disability index. J Rehabil Med. 2002 Nov;34(6):284-7. doi: 10.1080/165019702760390383. PMID 12440803
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Derived] Siddiqui M, Akhter S, Baig AAM. Effects of autogenic and reciprocal inhibition techniques with conventional therapy in mechanical neck pain - a randomized control trial. BMC Musculoskelet Disord. 2022 Jul 25;23(1):704. doi: 10.1186/s12891-022-05668-0. PMID 35879756